CLINICAL TRIAL: NCT05410600
Title: Smart Trainer Arm Ergometry Exercise Training in Individuals Post-Stroke (RERC on Technologies to Promote Exercise and Health Among People With Disabilities)
Brief Title: Smart Trainer Arm Ergometry Exercise Training in Individuals Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Rimmer, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300009387; 90REGE000 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2022-05-19; First posted 2022-06-08 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Exercise; Arm ergometer; Virtual environment; Disability
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Ergometer Smart Trainer Cycling (Experimental): Participants will participate in an 8-week exercise training program using the smart trainer.
  Interventions: Other: Arm ergometer smart trainer cycling program

INTERVENTIONS:
Other: Arm ergometer smart trainer cycling program — Arm ergometer exercise training using the smart trainer.

SUMMARY:
The smart trainer ergometer is comprised of an ergometer with foot and hand pedals, and a visual display in front of the user that can show a variety of scenic pathways. The purpose of this study is to examine changes in power output, oxygen consumption, cognitive function, and quality of life after 8 weeks of smart trainer arm ergometry exercise training among individuals with post-stroke limb impairment.

DETAILED DESCRIPTION:
Individuals with physical disabilities show much lower rates of exercise participation than their able-bodied peers. Much of the reason for the low rates of activity among this population comes from the presence of barriers. Lack of motivation, lack of transportation, lack of accessible facilities and equipment, and cost are all factors that discourage exercise participation among those with disabilities. Based on these factors, there is a need for accessible enjoyable exercise options for people with physical disabilities. The smart trainer ergometer (also known as the Advanced Virtual Exercise Environment Device) is comprised of an ergometer with foot and hand pedals, and a visual display in front of the user that can show a variety of scenic pathways.

In our previous protocol (IRB-300001384) we explored the power output curves of people post stroke compared with non-impaired individuals during one arm versus two arm cycling exercise using the smart trainer arm ergometer. The work demonstrated the potential benefit of interactive exercise for those with physical disabilities. The purpose of this study is to examine changes in power output, oxygen consumption, cognitive function, and quality of life after 8 weeks of smart trainer arm ergometry exercise training among individuals who have a stroke-based limb impairment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females post-stroke
* Age 40-70 years
* Able to use both arms during arm cycling exercise (i.e., able to complete the 10 revolution pre-test)

Exclusion Criteria:

* Younger than 40 and older than 70 years
* No movement in one arm or have an injury that prevents safe use of one arm during exercise
* Unable to complete the 10 revolution pre-test
* Unstable cardiovascular conditions
* Unable to understand study directions

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Consumption from Baseline to end of Week 8 | 8 weeks
  Oxygen consumption (VO2) as measured during a graded exercise test using a portable metabolic system

SECONDARY OUTCOMES:
Stroke Severity from Baseline to end of Week 8 | 8 weeks
  NIH Stroke Scale Test. Scores range from 0 to 42. A higher score indicates greater functional impairment.
Cognitive Function from Baseline to end of Week 8 | 8 weeks
  Mini-Mental State Exam. Scores range from 0 to 30, scores of 26 or higher indicate normal cognitive function
Quality of Life from Baseline to end of Week 8 | 8 weeks
  Stroke Impact Scale. Scores range from 0 to 100, with higher scores indicating higher quality of life.
Fatigue Severity from Baseline to end of Week 8 | 8 weeks
  Fatigue Severity Scale. Scores range from 9 to 63, with higher scores indicating greater fatigue severity.
Grip Strength from Baseline to end of Week 8 | 8 weeks
  Grip strength as measured using a hand dynamometer
Usability of the Smart Trainer at the end of Week 8 | 8 weeks
  System Usability Scale. Scores range from 0 to 100. Scores above 68 indicate above average usability. Scores below 68 point to issues with the design that need to be researched and resolved, while scores higher than 68 indicate the need for minor improvements to the design.
Participant feedback regarding the Smart Trainer Program at the end of Week 8 | 8 weeks
  Semi-structured interview to capture participant feedback regarding the smart trainer exercise training program and ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: James H Rimmer, PhD, Principal Investigator — UAB School of Health Professions
Locations (1):
- WHARF, Homewood, Alabama, United States